CLINICAL TRIAL: NCT03880838
Title: Evaluation of a Letter Intervention Among At-risk Adults Promoting a Plant-based Diet Using a Combination of Provider Testimonials, the Forks Over Knives Documentary, and Commitment- or Prevention-focused Behavioral Nudges
Brief Title: Evaluation of a Letter Intervention Promoting a Plant-based Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Geisinger Clinic
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2019-0179
Record Dates: First submitted 2019-03-14; First posted 2019-03-19 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus; Obesity
Keywords: Plant-based diet; Behavioral nudge; Mail distribution; Randomized controlled trial; Insurance claims; Chronic disease; Letter-based intervention; Health behaviors; Prevention focus; Loss framing; Commitment; Provider testimonial
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Obesity; Chronic Disease; Health Behavior

STUDY DESIGN:
Intervention Model Description: One group of participants will not be contacted at all (n = 6200). One group will only received a letter promoting a plant-based diet (n = 2200). Twelve groups (n = 550 for each group) will receive the letter promoting a plant-based diet, along with the Forks Over Knives documentary. The documentary will be delivered through 3 different methods, and the accompanying letter will contain 4 different combinations of behavioral nudges.
  * 1 primary control group (no contact)
  * 1 group contacted by letter
  * 3 groups (documentary distribution: online link, DVD, online link + DVD) x 4 groups (behavioral nudges in the letter: no nudge, commitment nudge, prevention nudge, commitment and prevention nudges)
  Note: The control group size is an estimate of number of participants who match the eligibility criteria but were not randomly assigned to an experimental group.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants, care providers, and outcomes assessors will not know the participant's arm. Insurance claims data and medical health records will be used (after all identifying information is removed).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- No contact control (No Intervention): Participants are not contacted.
- Letter (Experimental): Participants are only contacted through a letter with a personal testimonial.
  Interventions: Behavioral: Personal testimonial
- Link and no nudge (Experimental): Participants are sent the Forks Over Knives documentary online link and a letter with a personal testimonial and no nudges.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary
- Link and commitment nudge (Experimental): Participants are sent the Forks Over Knives documentary online link and a letter with a personal testimonial and a commitment nudge.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary; Behavioral: Commitment nudge
- Link and prevention nudge (Experimental): Participants are sent the Forks Over Knives documentary online link and a letter with a personal testimonial and a prevention nudge.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary; Behavioral: Prevention nudge
- Link and both nudges (Experimental): Participants are sent the Forks Over Knives documentary online link and a letter with a personal testimonial and both commitment and prevention nudges.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary; Behavioral: Commitment nudge; Behavioral: Prevention nudge
- DVD and no nudge (Experimental): Participants are sent the Forks Over Knives documentary DVD and a letter with a personal testimonial and no behavioral nudges.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary
- DVD and commitment nudge (Experimental): Participants are sent the Forks Over Knives documentary DVD and a letter with a personal testimonial and a commitment nudge.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary; Behavioral: Commitment nudge
- DVD and prevention nudge (Experimental): Participants are sent the Forks Over Knives documentary DVD and a letter with a personal testimonial and a prevention nudge.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary; Behavioral: Prevention nudge
- DVD and both nudges (Experimental): Participants are sent the Forks Over Knives documentary DVD and a letter with a personal testimonial and both commitment and prevention nudges.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary; Behavioral: Commitment nudge; Behavioral: Prevention nudge
- Link and DVD and no nudge (Experimental): Participants are sent the Forks Over Knives documentary online link and DVD and a letter with a personal testimonial and no behavioral nudges.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary
- Link and DVD and commitment nudge (Experimental): Participants are sent the Forks Over Knives documentary online link and DVD and a letter with a personal testimonial and a commitment nudge.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary; Behavioral: Commitment nudge
- Link and DVD and prevention nudge (Experimental): Participants are sent the Forks Over Knives documentary online link and DVD and a letter with a personal testimonial and a prevention nudge.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary; Behavioral: Prevention nudge
- Link and DVD and both nudges (Experimental): Participants are sent the Forks Over Knives documentary online link and DVD and a letter with a personal testimonial and both commitment and prevention nudges.
  Interventions: Behavioral: Personal testimonial; Behavioral: Forks Over Knives Documentary; Behavioral: Commitment nudge; Behavioral: Prevention nudge

INTERVENTIONS:
Behavioral: Personal testimonial — Participants will receive a letter promoting a plant-based diet. This letter will feature a personal testimonial about the benefits of a plant-based diet. Presenting this information to participants might encourage them to make behavioral changes to improve their health.
  Arms: DVD and both nudges; DVD and commitment nudge; DVD and no nudge; DVD and prevention nudge; Letter; Link and DVD and both nudges; Link and DVD and commitment nudge; Link and DVD and no nudge; Link and DVD and prevention nudge; Link and both nudges; Link and commitment nudge; Link and no nudge; Link and prevention nudge
Behavioral: Forks Over Knives Documentary — Participants will be mailed the documentary Forks Over Knives, which provides scientific arguments promoting a plant-based and whole foods diet. The behavioral effect of this documentary comes from watching the documentary and potentially choosing to order a free cookbook (participants are given this opportunity in the letter accompanying the documentary). The effect of the diet itself is not a central part of the intervention, as people can choose to adopt or not adopt any part of the diet.
  Arms: DVD and both nudges; DVD and commitment nudge; DVD and no nudge; DVD and prevention nudge; Link and DVD and both nudges; Link and DVD and commitment nudge; Link and DVD and no nudge; Link and DVD and prevention nudge; Link and both nudges; Link and commitment nudge; Link and no nudge; Link and prevention nudge
Behavioral: Commitment nudge — At the end of the letter promoting a plant-based diet, participants will be asked to write dates and personal signatures committing to watching the documentary. They will be asked to mail back this written commitment. Stating one's intentions to implement certain behavior is meant to increase the likelihood of follow-up behavior. This request might nudge more people to watch the documentary and make some behavioral changes to prevent negative health outcomes.
  Arms: DVD and both nudges; DVD and commitment nudge; Link and DVD and both nudges; Link and DVD and commitment nudge; Link and both nudges; Link and commitment nudge
Behavioral: Prevention nudge — As part of the letter promoting a plant-based diet, one paragraph will describe the risks of not taking action. This phrasing reframes the status quo as contributing to future loss (e.g., costs of medication and operations). In effect, the letter encourages participants to focus on preventing this loss by taking action. This additional text might nudge more people to watch the documentary and make some behavioral changes to prevent negative health outcomes.
  Arms: DVD and both nudges; DVD and prevention nudge; Link and DVD and both nudges; Link and DVD and prevention nudge; Link and both nudges; Link and prevention nudge

SUMMARY:
The researchers' mission is to promote healthier eating behavior and to reduce costs associated with healthcare. The purpose of this study is to evaluate the effects of mailing randomly selected participants a letter promoting a plant-based diet. Depending on the experimental condition, participants may additionally receive a free documentary, Forks Over Knives, and they may also get letters which use commitment- or prevention-focused messages to encourage watching the documentary and changing their eating behavior. The researchers hypothesize that receiving the documentary will be associated with lower insurance claims and improved health outcomes one and two years later. The researchers also hypothesize that using either commitment- or prevention-focused messages will also contribute to lower insurance claims and improved health outcomes compared to experimental conditions where materials did not include these messages. This study will help the researchers design evidence-supported programs that can improve people's health.

DETAILED DESCRIPTION:
Note that participant selection and assignment will be done at the level of the household, but analysis of outcomes will include individual-level analysis. This analytic decision was made because the researchers assume that the intervention may potentially affect other members of the household. While one person in a household will be selected for matching the eligibility criteria, the mailed materials will be addressed to all adult members of the household (defined as adults 18+ who are the spouse or child of the selected member) who are members of the Geisinger Health Plan. Outcome data will be pulled from all adult members of the household who have data through the Geisinger Health Plan.

The researchers will analyze the data using standard survey research analyses methods, including computing bivariate correlations, using general linear models, using non-parametric models for non-normally distributed insurance data, and entering variables as independent predictors in regression models to attempt to predict desired outcomes. The researchers will also use multilevel models to account for household- and individual-level data. The analysis of primary outcomes will focus on data one year after the intervention begins. Follow-up analysis on secondary outcomes will be conducted two years after the intervention begins. The researchers will conduct separate analyses of the selected participant (i.e., the individual who met the eligibility criteria) and other members of that participant's household. This will test whether there are any spillover effects of the intervention to other people in the household.

For clarity in this record, any discussion of sample size and participants refers to households, as this is the primary level for participant selection and assignment.

ELIGIBILITY:
Inclusion Criteria:

* Has two out of the three following conditions:

  * Body mass index over 30
  * Diagnosis of type 2 diabetes (specifically with at least one medication)
  * Diagnosis of cardiovascular disease
* Has health insurance through Geisinger Health Plan (is an active member with a full 12-month enrollment in the previous year) under one of the following categories:

  * Medicare with required primary care provider
  * Medicaid
  * Individual policy under the Affordable Care Act
* Has visited their primary care provider in the past 12 months

Exclusion Criteria:

* Is institutionalized
* Has active cancer, cirrhosis, renal failure, dementia, or active psychosis
* Is in the same household as another selected participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11234 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Program Director; Henri Carlo Y Santos, PhD, Study Director — Post-doctoral Fellow; Christopher Chabris, PhD, Study Director — Professor; Michelle N Meyer, PhD, JD, Study Director — Assistant Professor; Allison Hess, BS, Study Director — Vice President
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include preregistered hypotheses, analysis plan and code, and the essential data needed to replicate the analysis that yielded reported findings.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available upon publication and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

REFERENCES:
- [Background] Milkman KL, Beshears J, Choi JJ, Laibson D, Madrian BC. Using implementation intentions prompts to enhance influenza vaccination rates. Proc Natl Acad Sci U S A. 2011 Jun 28;108(26):10415-20. doi: 10.1073/pnas.1103170108. Epub 2011 Jun 13. PMID 21670283
- [Background] Tversky A, Kahneman D. The framing of decisions and the psychology of choice. Science. 1981 Jan 30;211(4481):453-8. doi: 10.1126/science.7455683.
- See also: The trailer for the Forks Over Knives Documentary that will be sent for free to participants in the relevant arms — https://www.forksoverknives.com/the-film

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The list of eligible participants was randomized before mail was sent (or not sent for no contact control group).
Groups:
- No Contact Control: Participants were not contacted.
- Letter: Participants were only contacted through a letter with a personal testimonial.
- Link and no Nudge: Participants were sent the Forks Over Knives documentary online link and a letter with a personal testimonial and no nudges.
- Link and Commitment Nudge: Participants were sent the Forks Over Knives documentary online link and a letter with a personal testimonial and a commitment nudge.
- Link and Prevention Nudge: Participants were sent the Forks Over Knives documentary online link and a letter with a personal testimonial and a prevention nudge.
- Link and Both Nudges: Participants were sent the Forks Over Knives documentary online link and a letter with a personal testimonial and both commitment and prevention nudges.
- DVD and no Nudge: Participants were sent the Forks Over Knives documentary DVD and a letter with a personal testimonial and no behavioral nudges.
- DVD and Commitment Nudge: Participants were sent the Forks Over Knives documentary DVD and a letter with a personal testimonial and a commitment nudge.
- DVD and Prevention Nudge: Participants were sent the Forks Over Knives documentary DVD and a letter with a personal testimonial and a prevention nudge.
- DVD and Both Nudges: Participants were sent the Forks Over Knives documentary DVD and a letter with a personal testimonial and both commitment and prevention nudges.
- Link and DVD and no Nudge: Participants were sent the Forks Over Knives documentary online link and DVD and a letter with a personal testimonial and no behavioral nudges.
- Link and DVD and Commitment Nudge: Participants were sent the Forks Over Knives documentary online link and DVD and a letter with a personal testimonial and a commitment nudge.
- Link and DVD and Prevention Nudge: Participants were sent the Forks Over Knives documentary online link and DVD and a letter with a personal testimonial and a prevention nudge.
- Link and DVD and Both Nudges: Participants were sent the Forks Over Knives documentary online link and DVD and a letter with a personal testimonial and both commitment and prevention nudges.
Period: Overall Study
Arm/Group | No Contact Control | Letter | Link and no Nudge | Link and Commitment Nudge | Link and Prevention Nudge | Link and Both Nudges | DVD and no Nudge | DVD and Commitment Nudge | DVD and Prevention Nudge | DVD and Both Nudges | Link and DVD and no Nudge | Link and DVD and Commitment Nudge | Link and DVD and Prevention Nudge | Link and DVD and Both Nudges
Started | 2434 | 2200 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550
Completed | 2434 | 2200 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only data related to mailing or the outcomes were provided for this analysis. No demographic or other baseline data were analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Contact Control | Letter | Link and no Nudge | Link and Commitment Nudge | Link and Prevention Nudge | Link and Both Nudges | DVD and no Nudge | DVD and Commitment Nudge | DVD and Prevention Nudge | DVD and Both Nudges | Link and DVD and no Nudge | Link and DVD and Commitment Nudge | Link and DVD and Prevention Nudge | Link and DVD and Both Nudges | Total
Number analyzed (Participants) | 2434 | 2200 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 11234
Age, Categorical [Count of Participants; unit: Participants] — Population: Data was not collected.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data was not collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2434 | 2200 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 550 | 11234

OUTCOME MEASURES:

1. Primary Outcome: Medical Cost in US Dollars From One Year Before to One Year After Intervention
Description: Total annual amount of medical and pharmacy costs (sum) as reported by Geisinger Health Plan. General linear models are used to model change between the data from the year before the intervention and the data from one year after intervention. Lower costs is the desirable outcome.
Time Frame: 2 years
Population: Number of participants analyzed was based on the number of baseline (2019) records with no missing data for this outcome.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | No Contact Control | Letter | Link and no Nudge | Link and Commitment Nudge | Link and Prevention Nudge | Link and Both Nudges | DVD and no Nudge | DVD and Commitment Nudge | DVD and Prevention Nudge | DVD and Both Nudges | Link and DVD and no Nudge | Link and DVD and Commitment Nudge | Link and DVD and Prevention Nudge | Link and DVD and Both Nudges
Number analyzed (Participants) | 1997 | 1849 | 434 | 466 | 459 | 447 | 453 | 453 | 458 | 458 | 472 | 454 | 451 | 457
dollars
  2019 | 6123.39 (9447.33) | 5863.82 (11818.81) | 5901.99 (11124.11) | 5630.26 (7461.85) | 6427.50 (9412.89) | 6343.24 (9206.43) | 6270.08 (9647.26) | 6336.36 (9452.46) | 6129.37 (10795.32) | 5542.03 (7632.87) | 6681.14 (10538.91) | 6850.98 (11812.93) | 6202.43 (8509.40) | 5305.93 (6743.15)
  2020 | 6101.54 (10076.51) | 6309.49 (13727.90) | 5754.70 (11157.93) | 5932.12 (8279.96) | 6078.06 (9847.06) | 7047.98 (14827.87) | 6284.85 (10203.78) | 6772.89 (10159.36) | 6709.80 (14548.68) | 5753.38 (7720.93) | 6723.81 (13785.71) | 6795.82 (12895.57) | 6275.88 (9067.47) | 5260.87 (6808.98)

2. Primary Outcome: Number of Visits From One Year Before to One Year After Intervention
Description: Total number of primary care physician and specialist visits (sum) as reported by Geisinger Health Plan. General linear models are used to model change between the data from the year before the intervention and the data from one year after intervention. Fewer visits is the desirable outcome.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | No Contact Control | Letter | Link and no Nudge | Link and Commitment Nudge | Link and Prevention Nudge | Link and Both Nudges | DVD and no Nudge | DVD and Commitment Nudge | DVD and Prevention Nudge | DVD and Both Nudges | Link and DVD and no Nudge | Link and DVD and Commitment Nudge | Link and DVD and Prevention Nudge | Link and DVD and Both Nudges
Number analyzed (Participants) | 1997 | 1849 | 434 | 466 | 459 | 447 | 453 | 453 | 458 | 458 | 472 | 454 | 451 | 457
visits
  2019 | 5.59 (6.31) | 5.57 (6.12) | 5.17 (5.91) | 5.66 (6.76) | 5.69 (6.12) | 5.77 (5.84) | 5.69 (5.49) | 5.43 (6.08) | 5.60 (6.74) | 5.88 (6.13) | 5.71 (6.25) | 5.59 (7.87) | 5.53 (5.89) | 5.26 (6.15)
  2020 | 4.77 (5.65) | 4.80 (5.56) | 4.26 (5.30) | 4.88 (5.78) | 4.89 (5.52) | 5.13 (5.36) | 4.82 (5.29) | 4.51 (5.31) | 4.49 (5.49) | 5.27 (5.80) | 5.15 (5.85) | 4.69 (6.24) | 4.63 (5.18) | 4.34 (5.06)

3. Primary Outcome: Number of Prescriptions From One Year Before to One Year After Intervention
Description: Total number of prescriptions (fills) as reported by Geisinger Health Plan. General linear models are used to model change between the data from the year before the intervention and the data from one year after intervention. Fewer prescriptions is the desirable outcome.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: prescriptions
Arm/Group | No Contact Control | Letter | Link and no Nudge | Link and Commitment Nudge | Link and Prevention Nudge | Link and Both Nudges | DVD and no Nudge | DVD and Commitment Nudge | DVD and Prevention Nudge | DVD and Both Nudges | Link and DVD and no Nudge | Link and DVD and Commitment Nudge | Link and DVD and Prevention Nudge | Link and DVD and Both Nudges
Number analyzed (Participants) | 1735 | 1580 | 381 | 403 | 391 | 404 | 403 | 395 | 399 | 411 | 413 | 395 | 382 | 399
prescriptions
  2019 | 48.96 (49.89) | 48.02 (48.47) | 47.44 (49.70) | 50.85 (46.95) | 50.50 (46.08) | 49.66 (43.44) | 49.14 (54.80) | 52.71 (53.75) | 48.66 (43.52) | 49.34 (48.53) | 48.82 (51.30) | 50.02 (49.10) | 50.26 (49.83) | 43.81 (44.03)
  2020 | 29.87 (47.45) | 26.82 (31.06) | 29.09 (62.85) | 29.86 (32.26) | 29.32 (33.00) | 30.35 (32.78) | 28.05 (32.78) | 30.24 (51.07) | 30.32 (35.34) | 31.70 (34.24) | 29.83 (36.16) | 27.83 (29.20) | 31.69 (36.72) | 27.30 (32.97)

4. Primary Outcome: Number of Unique Prescribed Medication From One Year Before to One Year After Intervention
Description: Total number of unique prescribed medication in the past year as reported by Geisinger Health Plan. General linear models are used to model change between the data from the year before the intervention and the data from one year after intervention. Less unique prescribed medication is the desirable outcome.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: prescriptions
Arm/Group | No Contact Control | Letter | Link and no Nudge | Link and Commitment Nudge | Link and Prevention Nudge | Link and Both Nudges | DVD and no Nudge | DVD and Commitment Nudge | DVD and Prevention Nudge | DVD and Both Nudges | Link and DVD and no Nudge | Link and DVD and Commitment Nudge | Link and DVD and Prevention Nudge | Link and DVD and Both Nudges
Number analyzed (Participants) | 1735 | 1580 | 381 | 403 | 391 | 404 | 403 | 395 | 399 | 411 | 413 | 395 | 382 | 399
prescriptions
  2019 | 8.12 (6.08) | 8.15 (6.22) | 7.90 (6.08) | 8.50 (6.25) | 8.47 (6.29) | 8.48 (5.76) | 7.84 (6.18) | 8.77 (7.52) | 8.32 (6.11) | 8.39 (7.07) | 8.25 (6.17) | 8.45 (6.43) | 8.53 (6.63) | 7.50 (6.15)
  2020 | 5.92 (4.86) | 5.82 (5.05) | 5.80 (4.93) | 6.27 (5.28) | 6.00 (5.31) | 6.28 (5.36) | 5.70 (4.77) | 5.98 (6.18) | 6.13 (5.43) | 6.44 (5.99) | 6.28 (5.28) | 5.88 (4.68) | 6.39 (5.47) | 5.66 (4.96)

5. Primary Outcome: Body Mass Index From One Year Before to One Year After Intervention
Description: Taken from annual checkup with primary care provider. Computed from height (in meters) and weight (in kilograms) data with the formula kilograms/meters^2. General linear models are used to model change between the data from the year before the intervention and the data from one year after intervention. A body mass index between the range of 18.5 to 25 is the desirable outcome.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | No Contact Control | Letter | Link and no Nudge | Link and Commitment Nudge | Link and Prevention Nudge | Link and Both Nudges | DVD and no Nudge | DVD and Commitment Nudge | DVD and Prevention Nudge | DVD and Both Nudges | Link and DVD and no Nudge | Link and DVD and Commitment Nudge | Link and DVD and Prevention Nudge | Link and DVD and Both Nudges
Number analyzed (Participants) | 2206 | 2022 | 500 | 506 | 505 | 497 | 503 | 510 | 499 | 506 | 516 | 512 | 498 | 509
kg/m^2
  2019 | 36.44 (7.35) | 36.48 (7.72) | 36.46 (7.53) | 36.20 (7.81) | 37.26 (7.59) | 36.58 (7.67) | 36.83 (8.76) | 36.56 (7.93) | 36.48 (7.33) | 37.00 (8.16) | 36.12 (7.67) | 36.83 (7.87) | 36.68 (7.80) | 35.76 (7.05)
  2020 | 36.06 (7.44) | 36.05 (7.61) | 36.16 (7.67) | 36.18 (8.11) | 36.77 (7.72) | 36.19 (7.63) | 36.39 (8.42) | 35.96 (7.58) | 36.11 (7.72) | 36.77 (8.80) | 35.73 (7.66) | 36.42 (8.08) | 36.30 (7.92) | 35.30 (7.05)
Statistical Analysis 1: Comparison: Letter vs Link and no Nudge vs Link and Commitment Nudge vs Link and Prevention Nudge vs Link and Both Nudges vs DVD and no Nudge vs DVD and Commitment Nudge vs DVD and Prevention Nudge vs DVD and Both Nudges vs Link and DVD and no Nudge vs Link and DVD and Commitment Nudge vs Link and DVD and Prevention Nudge vs Link and DVD and Both Nudges; In this contrast, letter was compared against all other conditions (coded into one category and set as the reference group). The key outcome is the interaction between conditions and time (2019 as the reference group); Test type: Superiority; p = .391, Regression, Linear; Slope = -0.06, Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: No Contact Control vs Link and no Nudge vs Link and Commitment Nudge vs Link and Prevention Nudge vs Link and Both Nudges vs DVD and no Nudge vs DVD and Commitment Nudge vs DVD and Prevention Nudge vs DVD and Both Nudges vs Link and DVD and no Nudge vs Link and DVD and Commitment Nudge vs Link and DVD and Prevention Nudge vs Link and DVD and Both Nudges; In this contrast, no contact control was compared against all other conditions (coded into one category and set as the reference group). The key outcome is the interaction between conditions and time (2019 as the reference group); Test type: Superiority; p = .861, Regression, Linear; Slope = -0.01, Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Link and no Nudge vs Link and Prevention Nudge vs DVD and no Nudge vs DVD and Prevention Nudge vs Link and DVD and no Nudge vs Link and DVD and Prevention Nudge; In this contrast, prevention conditions (coded into one category) were compared against no nudge conditions (coded into one category and set as the reference group); Test type: Superiority; p = .835, Regression, Linear; Slope = -0.02, Standard Deviation 0.01
Statistical Analysis 4: Comparison: Link and no Nudge vs Link and Commitment Nudge vs DVD and no Nudge vs DVD and Commitment Nudge vs Link and DVD and no Nudge vs Link and DVD and Commitment Nudge; In this contrast, commitment conditions (coded into one category) were compared against no nudge conditions (coded into one category and set as the reference group); Test type: Superiority; p = .877, Regression, Linear; Slope = .02, Standard Error of Mean 0.01
Statistical Analysis 5: Comparison: Link and no Nudge vs Link and Both Nudges vs DVD and no Nudge vs DVD and Both Nudges vs Link and DVD and no Nudge vs Link and DVD and Both Nudges; In this contrast, both nudge conditions (coded into one category) were compared against no nudge conditions (coded into one category and set as the reference group); Test type: Superiority; p = .969, Regression, Logistic; Slope = .004, Standard Error of Mean 0.01
Statistical Analysis 6: Comparison: Letter vs Link and no Nudge vs DVD and no Nudge vs Link and DVD and no Nudge; In this contrast, no nudge conditions (coded into one category) were compared against the letter condition (set as the reference group); Test type: Superiority; p = .893, Regression, Linear; Slope = 0.06, Standard Error of Mean 0.09
Statistical Analysis 7: Comparison: Letter vs Link and Prevention Nudge vs DVD and Prevention Nudge vs Link and DVD and Prevention Nudge; In this contrast, In this contrast, prevention conditions (coded into one category) were compared against the letter condition (set as the reference group); Test type: Superiority; p = .689, Regression, Linear; Slope = 0.04, Standard Error of Mean 0.10
Statistical Analysis 8: Comparison: Letter vs Link and Commitment Nudge vs DVD and Commitment Nudge vs Link and DVD and Commitment Nudge; In this contrast, commitment conditions (coded into one category) were compared against the letter condition (set as the reference group); Test type: Superiority; p = .427, Regression, Linear; Slope = 0.08, Standard Error of Mean 0.10
Statistical Analysis 9: Comparison: Letter vs Link and Both Nudges vs DVD and Both Nudges vs Link and DVD and Both Nudges; In this contrast, both nudge conditions (coded into one category) were compared against the letter condition (set as the reference group); Test type: Superiority; p = .504, Regression, Linear; Slope = 0.07, Standard Error of Mean 0.10
Statistical Analysis 10: Comparison: No Contact Control vs Link and no Nudge vs DVD and no Nudge vs Link and DVD and no Nudge; In this contrast, no nudge conditions (coded into one category) were compared against the no contact condition (set as the reference group); Test type: Superiority; p = .893, Regression, Linear; Slope = 0.01, Standard Error of Mean 0.09
Statistical Analysis 11: Comparison: No Contact Control vs Link and Prevention Nudge vs DVD and Prevention Nudge vs Link and DVD and Prevention Nudge; In this contrast, prevention conditions (coded into one category) were compared against the no contact condition (set as the reference group); Test type: Superiority; p = .918, Regression, Linear; Slope = -0.01, Standard Error of Mean 0.09
Statistical Analysis 12: Comparison: No Contact Control vs Link and Commitment Nudge vs DVD and Commitment Nudge vs Link and DVD and Commitment Nudge; In this contrast, commitment conditions (coded into one category) were compared against the no contact condition (set as the reference group); Test type: Superiority; p = .755, Regression, Linear; Slope = 0.03, Standard Error of Mean 0.09
Statistical Analysis 13: Comparison: No Contact Control vs Link and Both Nudges vs DVD and Both Nudges vs Link and DVD and Both Nudges; In this contrast, both nudge conditions (coded into one category) were compared against the no contact condition (set as the reference group); Test type: Superiority; p = .858, Regression, Linear; Slope = 0.02, Standard Error of Mean 0.09

6. Primary Outcome: Systolic Blood Pressure From One Year Before to One Year After Intervention
Description: Taken from annual checkup with primary care provider. General linear models are used to model change between the data from the year before the intervention and the data from one year after intervention. Systolic blood pressure that is 120 millimeters of mercury (mmHg) or less is the desirable outcome.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | No Contact Control | Letter | Link and no Nudge | Link and Commitment Nudge | Link and Prevention Nudge | Link and Both Nudges | DVD and no Nudge | DVD and Commitment Nudge | DVD and Prevention Nudge | DVD and Both Nudges | Link and DVD and no Nudge | Link and DVD and Commitment Nudge | Link and DVD and Prevention Nudge | Link and DVD and Both Nudges
Number analyzed (Participants) | 2199 | 2018 | 498 | 505 | 502 | 494 | 503 | 510 | 497 | 506 | 514 | 512 | 497 | 506
mmHg
  2019 | 130.00 (17.57) | 129.88 (17.19) | 130.47 (17.97) | 131.4 (16.59) | 130.72 (17.33) | 129.27 (17.18) | 129.88 (16.97) | 127.98 (18.50) | 129.19 (17.03) | 131.46 (16.85) | 130.41 (17.32) | 129.59 (17.10) | 130.39 (17.17) | 129.29 (17.90)
  2020 | 129.50 (17.94) | 129.97 (18.31) | 130.57 (17.00) | 130.26 (19.08) | 129.91 (17.03) | 129.73 (18.17) | 129.53 (17.33) | 127.58 (18.13) | 129.37 (17.20) | 131.79 (17.33) | 129.63 (17.55) | 129.25 (18.01) | 129.90 (17.29) | 129.70 (17.67)
Statistical Analysis 1: Comparison: Letter vs Link and no Nudge vs Link and Commitment Nudge vs Link and Prevention Nudge vs Link and Both Nudges vs DVD and no Nudge vs DVD and Commitment Nudge vs DVD and Prevention Nudge vs DVD and Both Nudges vs Link and DVD and no Nudge vs Link and DVD and Commitment Nudge vs Link and DVD and Prevention Nudge vs Link and DVD and Both Nudges; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = .436, Regression, Linear; Slope = 0.36, Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: No Contact Control vs Link and no Nudge vs Link and Commitment Nudge vs Link and Prevention Nudge vs Link and Both Nudges vs DVD and no Nudge vs DVD and Commitment Nudge vs DVD and Prevention Nudge vs DVD and Both Nudges vs Link and DVD and no Nudge vs Link and DVD and Commitment Nudge vs Link and DVD and Prevention Nudge vs Link and DVD and Both Nudges; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = .539, Regression, Linear; Slope = -0.27, Standard Error of Mean 0.45
Statistical Analysis 3: Comparison: Link and no Nudge vs Link and Prevention Nudge vs DVD and no Nudge vs DVD and Prevention Nudge vs Link and DVD and no Nudge vs Link and DVD and Prevention Nudge; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = .994, Regression, Linear; Slope = 0.005, Standard Error of Mean 0.66
Statistical Analysis 4: Comparison: Link and no Nudge vs Link and Commitment Nudge vs DVD and no Nudge vs DVD and Commitment Nudge vs Link and DVD and no Nudge vs Link and DVD and Commitment Nudge; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = .700, Regression, Linear; Slope = -0.25, Standard Error of Mean 0.66
Statistical Analysis 5: Comparison: Link and no Nudge vs Link and Both Nudges vs DVD and no Nudge vs DVD and Both Nudges vs Link and DVD and no Nudge vs Link and DVD and Both Nudges; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = .258, Regression, Logistic; Slope = 0.75, Standard Error of Mean 0.66
Statistical Analysis 6: Comparison: Letter vs Link and no Nudge vs DVD and no Nudge vs Link and DVD and no Nudge; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = .428, Regression, Linear; Slope = -0.49, Standard Error of Mean 0.62
Statistical Analysis 7: Comparison: Letter vs Link and Prevention Nudge vs DVD and Prevention Nudge vs Link and DVD and Prevention Nudge; In this contrast, prevention conditions (coded into one category) were compared against the letter condition (set as the reference group); Test type: Superiority; p = .434, Regression, Linear; Slope = -0.48, Standard Error of Mean 0.62
Statistical Analysis 8: Comparison: Letter vs Link and Commitment Nudge vs DVD and Commitment Nudge vs Link and DVD and Commitment Nudge; [analysis description as in outcome 5, analysis 8]; Test type: Superiority; p = .228, Regression, Linear; Slope = -0.74, Standard Error of Mean 0.62
Statistical Analysis 9: Comparison: Letter vs Link and Both Nudges vs DVD and Both Nudges vs Link and DVD and Both Nudges; [analysis description as in outcome 5, analysis 9]; Test type: Superiority; p = .674, Regression, Linear; Slope = 0.26, Standard Error of Mean 0.62
Statistical Analysis 10: Comparison: No Contact Control vs Link and no Nudge vs DVD and no Nudge vs Link and DVD and no Nudge; [analysis description as in outcome 5, analysis 10]; Test type: Superiority; p = .799, Regression, Linear; Slope = 0.15, Standard Error of Mean 0.61
Statistical Analysis 11: Comparison: No Contact Control vs Link and Prevention Nudge vs DVD and Prevention Nudge vs Link and DVD and Prevention Nudge; [analysis description as in outcome 5, analysis 11]; Test type: Superiority; p = .794, Regression, Linear; Slope = 0.16, Standard Error of Mean 0.61
Statistical Analysis 12: Comparison: No Contact Control vs Link and Commitment Nudge vs DVD and Commitment Nudge vs Link and DVD and Commitment Nudge; [analysis description as in outcome 5, analysis 12]; Test type: Superiority; p = .871, Regression, Linear; Slope = -0.10, Standard Error of Mean 0.61
Statistical Analysis 13: Comparison: No Contact Control vs Link and Both Nudges vs DVD and Both Nudges vs Link and DVD and Both Nudges; [analysis description as in outcome 5, analysis 13]; Test type: Superiority; p = .139, Regression, Linear; Slope = 0.90, Standard Error of Mean 0.62

7. Primary Outcome: Diastolic Blood Pressure From One Year Before to One Year After Intervention
Description: Taken from annual checkup with primary care provider. General linear models are used to model change between the data from the year before the intervention and the data from one year after intervention. Systolic blood pressure that is 80 millimeters of mercury (mmHg) or less is the desirable outcome.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | No Contact Control | Letter | Link and no Nudge | Link and Commitment Nudge | Link and Prevention Nudge | Link and Both Nudges | DVD and no Nudge | DVD and Commitment Nudge | DVD and Prevention Nudge | DVD and Both Nudges | Link and DVD and no Nudge | Link and DVD and Commitment Nudge | Link and DVD and Prevention Nudge | Link and DVD and Both Nudges
Number analyzed (Participants) | 2199 | 2018 | 498 | 505 | 502 | 494 | 503 | 510 | 497 | 506 | 514 | 512 | 497 | 506
mmHg
  2019 | 72.91 (10.99) | 72.79 (10.91) | 72.95 (10.89) | 73.48 (10.09) | 72.93 (10.90) | 72.27 (10.40) | 72.57 (10.37) | 72.44 (11.13) | 72.80 (10.51) | 73.44 (10.78) | 73.26 (10.41) | 73.21 (10.51) | 73.11 (10.79) | 73.04 (10.68)
  2020 | 72.48 (11.07) | 72.90 (11.42) | 73.07 (10.96) | 73.10 (11.85) | 72.41 (10.85) | 72.65 (11.28) | 72.42 (11.38) | 72.77 (11.12) | 72.64 (11.34) | 73.88 (11.20) | 72.97 (10.79) | 72.47 (10.64) | 72.58 (10.79) | 72.79 (11.37)
Statistical Analysis 1: Comparison: Letter vs Link and no Nudge vs Link and Commitment Nudge vs Link and Prevention Nudge vs Link and Both Nudges vs DVD and no Nudge vs DVD and Commitment Nudge vs DVD and Prevention Nudge vs DVD and Both Nudges vs Link and DVD and no Nudge vs Link and DVD and Commitment Nudge vs Link and DVD and Prevention Nudge vs Link and DVD and Both Nudges; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = .357, Regression, Linear; Slope = 0.26, Standard Error of Mean 0.29
Statistical Analysis 2: Comparison: No Contact Control vs Link and no Nudge vs Link and Commitment Nudge vs Link and Prevention Nudge vs Link and Both Nudges vs DVD and no Nudge vs DVD and Commitment Nudge vs DVD and Prevention Nudge vs DVD and Both Nudges vs Link and DVD and no Nudge vs Link and DVD and Commitment Nudge vs Link and DVD and Prevention Nudge vs Link and DVD and Both Nudges; [analysis description as in outcome 5, analysis 2]; Test type: Superiority; p = .294, Regression, Linear; Slope = -0.29, Standard Error of Mean 0.28
Statistical Analysis 3: Comparison: Link and no Nudge vs Link and Prevention Nudge vs DVD and no Nudge vs DVD and Prevention Nudge vs Link and DVD and no Nudge vs Link and DVD and Prevention Nudge; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = .496, Regression, Linear; Slope = -0.28, Standard Error of Mean 0.40
Statistical Analysis 4: Comparison: Link and no Nudge vs Link and Commitment Nudge vs DVD and no Nudge vs DVD and Commitment Nudge vs Link and DVD and no Nudge vs Link and DVD and Commitment Nudge; [analysis description as in outcome 5, analysis 4]; Test type: Superiority; p = .722, Regression, Linear; Slope = -0.14, Standard Error of Mean 0.40
Statistical Analysis 5: Comparison: Link and no Nudge vs Link and Both Nudges vs DVD and no Nudge vs DVD and Both Nudges vs Link and DVD and no Nudge vs Link and DVD and Both Nudges; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = .445, Regression, Linear; Slope = 0.31, Standard Error of Mean 0.40
Statistical Analysis 6: Comparison: Letter vs Link and no Nudge vs DVD and no Nudge vs Link and DVD and no Nudge; [analysis description as in outcome 5, analysis 6]; Test type: Superiority; p = .531, Regression, Linear; Slope = -0.24, Standard Error of Mean 0.38
Statistical Analysis 7: Comparison: Letter vs Link and Prevention Nudge vs DVD and Prevention Nudge vs Link and DVD and Prevention Nudge; [analysis description as in outcome 6, analysis 7]; Test type: Superiority; p = .177, Regression, Linear; Slope = -0.51, Standard Error of Mean 0.38
Statistical Analysis 8: Comparison: Letter vs Link and Commitment Nudge vs DVD and Commitment Nudge vs Link and DVD and Commitment Nudge; [analysis description as in outcome 5, analysis 8]; Test type: Superiority; p = .314, Regression, Linear; Slope = -0.38, Standard Error of Mean 0.38
Statistical Analysis 9: Comparison: Letter vs Link and Both Nudges vs DVD and Both Nudges vs Link and DVD and Both Nudges; [analysis description as in outcome 5, analysis 9]; Test type: Superiority; p = .850, Regression, Linear; Slope = 0.07, Standard Error of Mean 0.38
Statistical Analysis 10: Comparison: No Contact Control vs Link and no Nudge vs DVD and no Nudge vs Link and DVD and no Nudge; [analysis description as in outcome 5, analysis 10]; Test type: Superiority; p = .391, Regression, Linear; Slope = 0.32, Standard Error of Mean 0.37
Statistical Analysis 11: Comparison: No Contact Control vs Link and Prevention Nudge vs DVD and Prevention Nudge vs Link and DVD and Prevention Nudge; [analysis description as in outcome 5, analysis 11]; Test type: Superiority; p = .906, Regression, Linear; Slope = 0.04, Standard Error of Mean 0.37
Statistical Analysis 12: Comparison: No Contact Control vs Link and Commitment Nudge vs DVD and Commitment Nudge vs Link and DVD and Commitment Nudge; [analysis description as in outcome 5, analysis 12]; Test type: Superiority; p = .635, Regression, Linear; Slope = 0.18, Standard Error of Mean 0.37
Statistical Analysis 13: Comparison: No Contact Control vs Link and Both Nudges vs DVD and Both Nudges vs Link and DVD and Both Nudges; [analysis description as in outcome 5, analysis 13]; Test type: Superiority; p = 0.093, Regression, Linear; Slope = 0.63, Standard Error of Mean 0.37

8. Secondary Outcome: Triglyceride Levels From One Year Before to One Year After Intervention
Description: One component of cholesterol, used if data is on health record. A triglyceride level of 150 milligrams per deciliter (mg/dl) or lower is the desirable outcome.
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2055-12

9. Secondary Outcome: Low-density Lipoprotein (LDL) Levels From One Year Before to One Year After Intervention
Description: One component of cholesterol, used if data is on health record. An LDL level of 100 milligrams per deciliter (mg/dl) or lower is the desirable outcome.
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2055-12

10. Secondary Outcome: Five Years Before to Two Years After Intervention in Depressed Mood and Anhedonia as Assessed by the Patient Health Questionnaire-2 (PHQ-2) (Extended Time Frame)
Description: Assesses depressed mood and anhedonia in the past two weeks; used if data is on health record. The sum of two items (each scored 0-3) is computed with a total score range of 0-6. A lower score is the desired outcome.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

11. Secondary Outcome: Hemoglobin A1c (hbA1c) From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: Test for diabetes, used if data is on health record. Percentage score reflects blood-glucose levels. An hbA1c level of 5.7% and below is the desirable outcome.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

12. Secondary Outcome: Low-density Lipoprotein/High-density Lipoprotein (LDL/HDL) Ratios From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: Computed as the ratio of LDL/HDL. An LDL/HDL ratio of 3 or less for men and 2.5 or less for women is the desirable outcome.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

13. Secondary Outcome: High-density Lipoprotein (HDL) Levels From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: One component of cholesterol, used if data is on health record. An HDL level of 60 milligrams per deciliter (mg/dl) or higher is the desirable outcome.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

14. Secondary Outcome: Low-density Lipoprotein (LDL) Levels From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: as for outcome 9
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

15. Secondary Outcome: Triglyceride Levels From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: as for outcome 8
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

16. Secondary Outcome: Diastolic Blood Pressure From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: Taken from annual checkup with primary care provider. Systolic blood pressure that is 80 millimeters of mercury (mmHg) or less is the desirable outcome.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

17. Secondary Outcome: Systolic Blood Pressure From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: Taken from annual checkup with primary care provider. Systolic blood pressure that is 120 millimeters of mercury (mmHg) or less is the desirable outcome.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

18. Secondary Outcome: Body Mass Index From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: Taken from annual checkup with primary care provider. Computed from height (in meters) and weight (in kilograms) data with the formula kilograms/meters^2. A body mass index between the range of 18.5 to 25 is the desirable outcome.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

19. Secondary Outcome: Number of Unique Prescribed Medication From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: Total number of unique prescribed medication in the past year as reported by Geisinger Health Plan. Less unique prescribed medication is the desirable outcome.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

20. Secondary Outcome: Number of Prescriptions From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: Total number of prescriptions (standard unit is prescription per number of days supplied) as reported by Geisinger Health Plan. Fewer prescriptions is the desirable outcome.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

21. Secondary Outcome: Number of Visits From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: Total number of primary care physician and specialist visits (sum) as reported by Geisinger Health Plan. Fewer visits is the desirable outcome.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

22. Secondary Outcome: Medical Cost in US Dollars From Five Years Before to Two Years After Intervention (Extended Time Frame)
Description: Total annual amount of medical and pharmacy costs (sum) as reported by Geisinger Health Plan. Lower costs is the desirable outcome.
Time Frame: 7 years
Reporting Status: Not Posted, anticipated posting 2055-12

23. Secondary Outcome: Values From One Year Before to One Year After Intervention of Depressed Mood and Anhedonia as Assessed by the Patient Health Questionnaire-2 (PHQ-2)
Description: Although originally listed as secondary, this outcome measure was intended to be exploratory. Due to the largely null pattern of results on the primary outcomes, it was decided to forgo additional analysis at this time.
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2055-12

24. Secondary Outcome: Hemoglobin A1c (hbA1c) From One Year Before to One Year After Intervention
Description: Test for diabetes, used if data is on health record. Percentage score reflects blood-glucose levels. An hbA1c level of 5.7% or lower is the desirable outcome.
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2055-12

25. Secondary Outcome: Low-density Lipoprotein/High-density Lipoprotein (LDL/HDL) Ratios From One Year Before to One Year After Intervention
Description: as for outcome 12
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2055-12

26. Secondary Outcome: High-density Lipoprotein (HDL) Levels From One Year Before to One Year After Intervention
Description: as for outcome 13
Time Frame: 2 years
Reporting Status: Not Posted, anticipated posting 2055-12

ADVERSE EVENTS:
Time Frame: We did not report a time frame as we did not actively collect adverse event data.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed. No adverse events were evaluated, as only data from the outcomes were gathered. Mortality was not a risk associated with participation in our study.
Arm/Group | No Contact Control | Letter | Link and no Nudge | Link and Commitment Nudge | Link and Prevention Nudge | Link and Both Nudges | DVD and no Nudge | DVD and Commitment Nudge | DVD and Prevention Nudge | DVD and Both Nudges | Link and DVD and no Nudge | Link and DVD and Commitment Nudge | Link and DVD and Prevention Nudge | Link and DVD and Both Nudges
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to limited data access, only information related to mailing and the outcomes were given to the researchers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT03880838/Prot_001.pdf
  • Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT03880838/SAP_000.pdf